CLINICAL TRIAL: NCT00952666
Title: Transrectal Ultrasound (TRUS) Imaging of the Prostate Gland and Neurovascular Bundles (NVB) During Robot-Assisted Laparoscopic Radical Prostatectomy (RALRP)
Brief Title: Transrectal Ultrasound Imaging of the Prostate Gland and Neurovascular Bundles During Robot-Assisted Laparoscopic Radical Prostatectomy
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The number of participants needed for this study has been met.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Misop Han, M.D., M.S., Johns Hopkins Medical Institutions
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00014120
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Last update posted 2010-09-13 (Estimated); Status verified 2009-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Transrectal Ultrasound Imaging of Prostate; Neurovascular Bundles; Robot Assisted Laparoscopic Radical Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Device (Experimental): Both the Robot-Assisted Laparoscopic Radical Prostatectomy (RALRP) and the Transrectal Ultrasound (TRUS) are common performed procedures, but are normally performed separately. In this proposed feasibility study, the procedures will be combined.
  Interventions: Device: TRUS-RALRP

INTERVENTIONS:
Device: TRUS-RALRP — During surgery, and part of this research study, the ultrasound probe (TRUS) will be placed in the rectum. Then, using the mechanical support arm to hold and adjust the probe we will take ultrasound images during a portion of the robotic LRP surgery. The ultrasound probe will then be removed, and we will complete the LRP surgery as we usually do. We expect this to add approximately 20 minutes to the regular surgery time; the maximum added time will be 30 minutes.
  Other Names: TRUS support arm with daVinci robot

SUMMARY:
Neurovascular bundle (NVB) contains capsular vessels to the prostate and cavernous nerves that provides the macroscopic landmark used during nerve-sparing radical prostatectomy. The preservation of NVB during radical prostatectomy improves postoperative recovery of potency and continence. However, the visualization of the NVB during radical prostatectomy can be challenging.

Recently, an attempt has been made to use a transrectal ultrasound (TRUS) imaging to delineate the anatomy of the prostate gland and NVB during laparoscopic radical prostatectomy. However, it is difficult to obtain a steady image of TRUS with an operator. The investigators plan to perform a feasibility study to obtain TRUS imaging of the prostate and NVB during robot-assisted laparoscopic radical prostatectomy (RALRP). The investigators plan to use a robot-assisted TRUS probe holder to gently manipulate the probe to obtain steady TRUS images that may aid in visualization and dissection of the NVB during RALRP.

DETAILED DESCRIPTION:
During surgery for prostate cancer, precise resection of the tumor-containing prostate gland and preservation of the neurovascular bundle (NVB) are critical in preventing tumor recurrence and potency preservation following surgery. However, due to the periprostatic connective tissues and bleeding, it is difficult to visualize NVB during surgery, even with surgical loupes or laparoscopic magnification.

Ultrasound (US) is commonly used in imaging the prostate during diagnostic and therapeutic procedures such as diagnostic biopsy. US image in addition to the classic laparoscopic imaging can potentially provide decreased surgical margins and improve the dissection of the NVB during laparoscopic radical prostatectomy (LRP) according to the study by the Cleveland Clinic group. In their study, an assistant manipulated the TRUS probe under the direction of the surgeon and held it in place as requested. At critical points of the surgery, the surgeon visualized the NVB on the Doppler-capable ultrasound monitor. The images, however, were difficult to interpret because the surgeon was not in direct control of the TRUS probe. In addition, it was challenging for surgeon to communicate with the assistant to obtain steady and useful image. Moreover, their study was performed exclusively in LRP without the daVinci® robot (Intuitive Surgical, Inc.), more commonly performed surgical approach for radical prostatectomy.

To overcome these obstacles in the study by Ukimura and al., we propose to use a mechanical support arm for holding and manipulating the TRUS probe during the daVinci® robot-assisted laparoscopic radical prostatectomy (robotic LRP)..

This application is for a feasibility study involving six patients. We will obtain TRUS images of the prostate and NVB during a robotic LRP procedure. These images will be acquired in the first part of the operation and performed with minimal interference to the operation. We will record and analyze the TRUS images to investigate the feasibility of using mechanical support arm for the TRUS probe. The proposed study is a proof of concept for a following protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for a Laparoscopic Radical Prostatectomy operation
* Patients must be between the ages of 35 and 75
* Patients must not have one of the above listed exclusion criteria
* Patients must be able to understand and willing to adhere to the study protocol

Exclusion Criteria:

* Patients less than 35 years of age and over 75 years of age
* Patients with previous rectal surgery
* Patients with anal stenosis that prevents the TRUS probe insertion
* Patients with extensive abdominal surgery
* Patients with inadequate bowel prep
* Patients who are unwilling or unable to sign informed consent
* Patients on anticoagulation medication (e.g., coumadin, lovenox, or heparin)

Ages: 35 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Misop Han, M.D., M.S., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States